CLINICAL TRIAL: NCT03727711
Title: "Transcutaneous Tibial Nerve Stimulation as a Conservative Treatment for Overactive Bladder Dysfunction -A Randomised Controlled Trial Comparing Home Versus Hospital Based Treatment"
Brief Title: TPTNS: Home vs Hospital Treatment for Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN15UR229
Record Dates: First submitted 2017-08-11; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Overactive Bladder; Detrusor, Overactive
Keywords: transcutaneous posterior tibial nerve stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home Treatment (Experimental): Participants will be taught home treatment with TPTNS - twice weekly, 30 minute sessions for 6 weeks
  Interventions: Other: TPTNS
- Hospital Treatment (Active Comparator): Participants will receive hospital treatment with TPTNS - twice weekly, 30 minute sessions for 6 weeks
  Interventions: Other: TPTNS

INTERVENTIONS:
Other: TPTNS — We will be comparing hospital treatment to TPTNS at home

SUMMARY:
Comparison of home versus hospital Transcutaneous Posterior Tibial Nerve Stimulation (TPTNS). TPTNS has been shown to be an effective treatment of overactive bladder in hospital. We aim to see if this effect is replicated at home.

80 patients will be recruited, 40 into each arm.

Inclusion criteria:

1. Women aged ≥18 years
2. Clinical diagnosis of Overactive Bladder (OAB)
3. Post-void residual urine volume of < 100ml
4. Able to do questionnaires
5. Able to consent and willing to participate

Exclusion Criteria

1. Cardiac pacemaker in situ
2. Leg ulcer/skin condition affecting both lower legs
3. Diagnosed peripheral vascular disease
4. Absent sensation at the electrode site
5. Current Urinary Tract Infection (UTI) - must be treated with appropriate antibiotics as per the unit protocol prior to commencing study
6. Pregnancy
7. Previous Percutaneous Tibial Nerve Stimulation (PTNS) /Sacral Nerve Stimulation (SNS) course
8. Previous intravesical botox treatment
9. Unable to complete questionnaires

TPTNS will be taught to the home group and delivered to the participants in the hospital group in individual appointments: 12 treatment sessions of 30 minutes duration, delivered twice weekly over a 6 week period. Two surface electrodes are applied to the right ankle. These electrodes are attached to an electrical stimulator, programmed to safely deliver electric pulses.

On completion of 6 sessions, all participants will be contacted and asked to do a Patient Global Impression of Improvement Scale (PGIIS) and Patient Perception of Bladder Condition (PPBC). After 12 sessions (the final treatment session) all participants will be reviewed by the investigators in the hospital and the outcome measures repeated. Participants receiving home treatment will be posted out a 3 day bladder diary to complete. At this point the participants receiving home treatment will return the machine. All participants will complete and return a 72-hour bladder diary and validated questionnaires routinely used at the study centre to measure lower urinary tract symptoms - The International Consultation of Incontinence Modular Questionnaire - Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) long form, the International Consultation of Incontinence Modular Questionnaire - Urinary Incontinence questionnaire (ICIQ-UI short-form. The Hospital Anxiety and Depression Scale (HADS) and the European Quality of Life - 5D Questionnaire (EQ-5D) will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women aged greater than or equal to 18 years

  2. Clinical diagnosis of OAB

  3. Post-void residual urine volume of < 100ml

  4. Able to do questionnaires

  5. Able to consent and willing to participate

Exclusion Criteria:

* 1. Cardiac pacemaker in situ

  2. Leg ulcer/skin condition affecting both lower legs

  3. Diagnosed peripheral vascular disease

  4. Absent sensation at the electrode site

  5. Current UTI - must be treated with appropriate antibiotics as per the unit protocol prior to commencing study

  6. Pregnancy

  7. Previous PTNS /SNS

  8. Previous intravesical botox treatment

  9. Unable to complete questionnaires

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-03-03 (Estimated); Study Completion 2019-08-04 (Estimated)

PRIMARY OUTCOMES:
Change in the International Consultation of Incontinence Modular - Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) Long Form Questionnaire total score | At 6 weeks (i.e. after the last TPTNS treatment) and at 12 weeks (i.e. 6 weeks after last the TPTNS treatment)
  The ICIQ-FLUTS Long Form is a patient-completed questionnaire for evaluating female lower urinary tract symptoms and impact on quality of life (QoL) - 18 questionnaire items are asked and summed to calculate total score. Total score range (0-69) - a higher score indicates a worse outcome. Bother scales are not incorporated in the overall score but indicate impact of individual symptoms for the patient .

SECONDARY OUTCOMES:
Change in number of urgency incontinence episodes recorded on 72 hour bladder diary. | At 6 weeks (i.e. after the last TPTNS treatment) and at 12 weeks (i.e. 6 weeks after last the TPTNS treatment)
  Patient Perception of Intensity of Urgency Severity (PPIUS) Scores on the bladder diary are recorded when a participant experiences incontinence (range 0-4): 0 indicates no urgency, 1-4 indicate urgency experienced (at increasing severity). Number of episodes of urge incontinence are identified and summed.
Change in individual urgency score on International Consultation of Incontinence Modular Questionnaire - Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) Long Form Questionnaire | At 6 weeks (i.e. after the last TPTNS treatment) and at 12 weeks (i.e. 6 weeks after last the TPTNS treatment)
  Change in numerical scores for Urgency. Scoring range on questionnaire (0-4) - a higher number indicates a worse outcome.
Change in individual frequency score on International Consultation of Incontinence Modular Questionnaire - Female Lower Urinary Tract Symptoms (ICIQ - FLUTS) Long Form Questionnaire | At 6 weeks (i.e. after the last TPTNS treatment) and at 12 weeks (i.e. 6 weeks after last the TPTNS treatment)
  Change in numerical score on the questionnaire. Scoring range on questionnaire (0-4) - a higher number indicates a worse outcome.
Change in individual nocturia score on International Consultation of Incontinence Modular Questionnaire - Female Lower Urinary Tract Symptoms (ICIQ - FLUTS) Long Form Questionnaire | At 6 weeks (i.e. after the last TPTNS treatment) and at 12 weeks (i.e. 6 weeks after last the TPTNS treatment)
  Change in numerical score on the questionnaire. Scoring range on questionnaire (0-4) - a higher number indicates a worse outcome.
Change in incontinence symptom severity | At 6 weeks (i.e. after the last TPTNS treatment) and at 12 weeks (i.e. 6 weeks after last the TPTNS treatment)
  Change in International Consultation of Incontinence Modular Questionnaire - Urinary Incontinence short-form (ICIQ-UI SF) numerical scores. Scoring range (0-21) - 4 subscales summed for overall score on questionnaire; a higher score indicates increased severity. Self-diagnostic item un-scored.
Change in Mean urgency perception scores recorded on 72 hour bladder diary • | At 6 weeks (i.e. after the last TPTNS treatment) and at 12 weeks (i.e. 6 weeks after last the TPTNS treatment)
  Change in Patient Perception of Intensity of Urgency Severity (PPIUS) Scores on the bladder diary. Range for PPIUS (0-4); a higher score indicates increased severity.
PGIS (Patient Global Impression of Improvement Scale) Score | At 6 weeks (i.e. after the last TPTNS treatment) and at 12 weeks (i.e. 6 weeks after last the TPTNS treatment)
  Change in numerical score on the questionnaire. Range (1-7); higher scores indicate least improvement.
Change in HADS (Hospital Anxiety and Depression) scores | At 6 weeks (i.e. after the last TPTNS treatment) and at 12 weeks (i.e. 6 weeks after last the TPTNS treatment)
  The HADS is a 14 item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Individual item score range (0-3) which are summed for total score. Total score range (0-21) for either Anxiety or Depression. Higher scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ciara M Daly, MB Bch BAO, Principal Investigator — Queen Elizabeth University Hospital Glasgow
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daly CME, Loi L, Booth J, Saidan D, Guerrero K, Tyagi V. Self-management of overactive bladder at home using transcutaneous tibial nerve stimulation: a qualitative study of women's experiences. BMC Womens Health. 2021 Oct 27;21(1):374. doi: 10.1186/s12905-021-01522-y. PMID 34706709